CLINICAL TRIAL: NCT01506778
Title: Using a Tenaculum Which is Actually Necessary for Endometrial Sampling Procedure by Pipelle.
Brief Title: Tenaculum in Endometrial Sampling Procedure
Acronym: Tenaculum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ümran Küçükgöz Güleç, Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CukurovaU
Record Dates: First submitted 2012-01-02; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Endometrium; Biopsy
Keywords: Endometrial Sampling Procedure; Likert Scala; Pipelle; Tenaculum; Visual Analog Pain Scala

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1(With Tenaculum) (Active Comparator): This group consisted of the patients whose had been applied tenaculum at cervix during the endometrial sampling procedure
  Interventions: Device: Tenaculum
- Group 2 (Without Tenaculum) (No Intervention): This group consisted of the patients whose had been not applied tenaculum during the endometrial sampling procedure.

INTERVENTIONS:
Device: Tenaculum — Single tooth tenaculum are use to the cervix for steady the cervix, straighten the cervicouterine angle and provide countertraction. Most of gynecological office procedure such as endometrial sampling procedure, hysterosalpingography, hysteroscopy, insertion of contraceptive intrauterine device, difficult intrauterine insemination or embryo transfer procedures often require the application of a tenaculum.
  Arms: Group 1(With Tenaculum)

SUMMARY:
Most of gynecological office procedure such as endometrial sampling procedure, hysterosalpingography, hysteroscopy, insertion of contraceptive intrauterine device, difficult intrauterine insemination or embryo transfer procedures often require the application of a single tooth tenaculum to the cervix for steady the cervix, straighten the cervicouterine angle and provide countertraction. However, grasping the cervix with a tenaculum can be a painful experience for the patient.A randomized controlled trial was conducted to evaluate using of tenaculum on pain perception of the patients and the procedure performance of the surgeons in endometrial sampling procedure(ESP) with pipelle.

DETAILED DESCRIPTION:
One hundred fifteen patients included for assessing pain perception and procedure performance during endometrial with pipelle. Patients were randomly assigned to one of two groups as Group 1( with tenaculum) and Group 2 (without tenaculum).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* The women has required endometrial sampling procedure in gynecology outpatients clinic.
* Who are capable understand the spoken words and describe the pain.

Exclusion Criteria:

* Stenotic cervical canal
* They had acute cervicitis
* Intense anxiety
* Need for coincident endocervical curettage
* Need for general anesthesia or local anesthetics
* The use of analgesic drug pre-procedure
* Known history of malignancy
* Uterine anomalies or leiomyomas that distort the cervical canal and cavity
* A history of failed office endometrial sampling
* Positive β-HCG test.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala for patient's pain perception | 5 second
  VAS performed four times each patient.

SECONDARY OUTCOMES:
Likert scala for procedure performance | 5 second
  Likert scaled one times by the physician.
Success rate as adequate sampling of endometrial tissue for histopathologic diagnosis. | 5-10 day

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Baris Guzel, Assist Prof Dr., Principal Investigator — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology; Aybala Kubat, MD, Principal Investigator — Şahinbey Goverment Hospital; Ghanim Khatib, MD, Principal Investigator — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology; Fatma Tuncay Ozgunen, Prof Dr., Principal Investigator — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology; Ibrahim Ferhat Urunsak, Assist Prof Dr., Principal Investigator — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology; Umran Kucukgoz Gulec, Assist Prof Dr., Study Director — Cukurova University Faculty of Medicine Department of Obstetrics and Gynecology
Locations (1):
- Cukurova University Faculty of Medicine, Adana, Turkey (Türkiye)